CLINICAL TRIAL: NCT02560012
Title: Targeting of Renal Cell Cancer With Specific Inhibitors: A Model for Selective Adaptive Medicine Based on Molecular Alterations
Brief Title: Personalized Targeted Inhibitors Treatment in Renal Cell Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Loss of laboratory performing molecular analysis
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Robert J Amato, Director and Professor, Department of Internal Medicine, Division of Oncology, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GU-14-102; HSC-14-0665 (Other: UTHealth Committee for Protection of Human Subjects)
Record Dates: First submitted 2015-09-17; First posted 2015-09-25 (Estimated); Results first posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-09

CONDITIONS: Carcinoma, Renal Cell
Keywords: Renal Cell Carcinoma; RCC; Personalized therapy; targeted inhibitors
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib; temsirolimus; Sorafenib; pazopanib; Everolimus; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Personalized therapy (Other): Subjects will receive one of the four first-line therapy agents based on their tumor's profile. The first-line agents are sunitinib, temsirolimus, sorafenib, or pazopanib. These are all routine drugs for RCC treatment and will be given at their approved doses and dosing schedules.
  Upon disease progression, subject's tumor(s) will be biopsied again to create another tumor profile. The second-line agents are everolimus or axitinib. Both of these are routine drugs for RCC treatment and will be given at their approved doses and dosing schedules.
  Interventions: Drug: Sunitinib; Drug: Temsirolimus; Drug: Sorafenib; Drug: Pazopanib; Drug: Everolimus; Drug: Axitinib

INTERVENTIONS:
Drug: Sunitinib — One 50-mg capsule taken orally once daily, on a schedule of 4 weeks on treatment followed by 2 weeks off
  Other Names: Sutent
Drug: Temsirolimus — 25 mg by an IV infusion over 30-60 minutes, once a week
  Other Names: Torisel
Drug: Sorafenib — 400 mg (2 tablets) orally twice daily without food
  Other Names: Nexavar
Drug: Pazopanib — 800 mg orally once a day without food, at least 1 hour before or 2 hours after a meal
  Other Names: Votrient
Drug: Everolimus — 10 mg orally once daily with or without food
  Other Names: Afinitor
Drug: Axitinib — 5 mg orally twice daily
  Other Names: Inlyta

SUMMARY:
This is for subjects with metastatic Renal Cell Cancer (RCC). There are four Food and Drug Administration (FDA) approved drugs for first-line therapy of Renal Cell Cancer (RCC) and two for second-line therapy. Each of these drugs targets a specific molecular pathway. At present oncologists select therapy based on current guidelines. There is a new method for trying to use biomarker information from the subject's tumor to select the best drug to treat the subject. This process is investigational, which is why this study is being done.

Biomarkers are genes, proteins and other molecules that affect how cancer cells grow, multiply, die and respond to other compounds in the body. These biomarkers build a tumor profile or "fingerprint" of the subject's tumor. A new focus in cancer care is personalized treatment, where doctors select a drug based on the subject's tumor's unique "fingerprint" which is more likely to be effective in fighting the tumor. Selecting the treatment the subject is more likely to respond to requires a thorough understanding of the relationship between biomarker and treatment effect. The PI wants to gather data to understand that relationship to help treat future cancer patients. The purpose of this study is to evaluate efficacy of treatments that are selected based on tumor profiles.

DETAILED DESCRIPTION:
This will be a prospective, one-arm, proof of concept study designed to evaluate the efficacy of algorithm-based allocation (based on genomic/proteomic profile) of first-line therapy in renal cell carcinoma (RCC).

After eligibility review, patients will receive one of the four first-line therapy agents based on their tumor's molecular profile as determined using fresh biopsy tissue from an accessible metastatic site. Upon disease progression, patients will then receive one of two second-line agents based on their tumor's molecular profile.

Because this is a proof-of-concept study, the sample size is based on feasibility of accrual. The clinic should be able to recruit 100 patients within a reasonable timeframe for the study. The number of patients receiving each drug will vary based on the frequency of molecular alterations in the population. Therefore, groups will not be compared with one another - the research goal is to determine whether the progression-free survival (PFS) for each drug is improved over the PFS reported in FDA approval trials for each drug when they are assigned based on molecular analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be included in the study only if they meet all of the following inclusion criteria:

  * Pathologically confirmed renal cell carcinoma.
  * No prior systemic and/or investigative therapy of any kind.

    * Patients with primary tumor in place are strongly encouraged to undergo nephrectomy prior to initiation of study agent.
    * Prior palliative radiotherapy to metastatic lesion(s) is permitted. Patient must have adequately recovered from the acute toxicities of this treatment.
    * All major surgery of any type and/or radiotherapy must be completed at least 4 weeks prior to registration.
  * Must have progressive metastatic disease
  * ECOG performance status ≤2
  * Women of childbearing potential and male patients must use acceptable methods of contraception-tubal ligation, vasectomy, barrier contraceptive with spermicide-while on study and for 3 months after the last dose of study therapy. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study.
  * Age ≥18 years
  * Required Initial Laboratory Values:

    * Granulocytes ≥1,500/µL
    * Platelet Count ≥100,000/µL
    * Hemoglobin ≥9 g/dL
    * AST/ALT ≤ 2.5 times the upper limit of normal (ULN)
    * Alk. Phos.≤ 2.5 x ULN
    * Serum bilirubin ≤ 1.5 x ULN
    * Amylase/Lipase within normal range
    * Urinalysis≤ 1+ protein
    * T3T4 TSH - within normal range
    * Pregnancy test for women - Negative
    * Serum creatinine ≤ 1.5 x ULN
    * Electrocardiogram (ECG) - no active ischemia
    * Echocardiogram ejection fraction ≥40%
    * Pulmonary function tests
    * Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
  * Signed informed consent prior to the performance of any study-specific procedures

Exclusion Criteria:

* Ongoing hemoptysis, or cerebrovascular accident within 12 months prior to study entry, or peripheral vascular disease with claudication occurring upon walking less than one city block, or history of clinically significant bleeding.
* Deep venous thrombosis or pulmonary embolus within 12 months prior to study entry and no ongoing need for full-dose oral or parenteral anticoagulation. For maintenance of catheter patency daily prophylactic aspirin or low-dose coumadin (1-2 mg) is allowed.
* Evidence of current central nervous system (CNS) metastases. All patients must undergo a CT scan of the brain (with contrast, if possible) within 42 days prior to registration. Any imaging abnormality indicative of active CNS metastases will exclude the patient from the study.
* Significant cardiovascular disease defined as congestive heart failure (New York Heart Association Class II, II or IV) angina pectoris requiring nitrate therapy, or recent myocardial infarction (within the preceding 6 months prior to study entry).
* Uncontrolled hypertension (defined as blood pressure of ≥160 mmHg systolic and/or ≥90 mmHg diastolic on medication). Document over 48 hours with minimum of 3 readings.
* Ongoing requirement for systemic corticosteroid therapy (except replacement therapy for adrenal insufficiency) or other immunosuppressants are not permitted. Topical and/or inhaled steroids are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2017-07-27 (Actual); Study Completion 2017-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Amato, DO, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- UTHealth Memorial Hermann Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One enrolled patient's tumor did not have a genomic profile completed as next-generation sequencing was not done. Both proteomics and genomics assessments were required so patient was excluded.
Groups:
- Personalized Therapy: Participants will receive one of four first-line therapy agents based on their tumor's profile. First-line agents are sunitinib, temsirolimus, sorafenib, or pazopanib. These are all routine drugs for RCC treatment and will be given at their approved doses and dosing schedules.
  Upon disease progression, participant's tumor will be biopsied again to create another tumor profile. The second-line agents are everolimus or axitinib. Both of these are routine drugs for RCC treatment and will be given at their approved doses and dosing schedules.
  Sunitinib: One 50-mg capsule taken orally once daily, on a schedule of 4 weeks on treatment followed by 2 weeks off
  Temsirolimus: 25 mg by an IV infusion over 30-60 minutes, once a week
  Sorafenib: 400 mg (2 tablets) orally twice daily without food
  Pazopanib: 800 mg orally once a day without food, at least 1 hour before or 2 hours after a meal
  Everolimus: 10 mg orally once daily with or without food
  Axitinib: 5 mg orally twice
Period: Overall Study
Arm/Group | Personalized Therapy
Started | 3
Completed | 1
Not Completed | 2
Not completed — Study Terminated | 2

BASELINE CHARACTERISTICS:
Arm/Group | Personalized Therapy
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: years] | 65 [46 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3
Eastern Cooperative Oncology Group Performance Status (ECOG) [Count of Participants; unit: Participants]
  0-Fully active, pre-disease performance | 3
  1-No strenuous activity, ambulatory, light work | 0
  2-Ambulatory, selfcare, unable to work | 0
  3-Limited selfcare, confined to bed/chair > 50% | 0
  4-Completely disabled, no selfcare, bed/chair 100% | 0
  5-Dead | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Progressed
Description: The PFS is defined as the time elapsed between treatment initiation and tumor progression or death from any cause, with censoring of patients who are lost to follow-up. Progression is defined using the Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1): " At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression)."
Time Frame: From date of enrollment until the date of first documented progression, date of death from any cause, or date that the study was stopped, whichever came first, an average of 16 months
Population: All participants who received personalized therapy (sunitinib, temsirolimus, sorafenib, or pazopanib) based on their tumor's profile.
Measure: Count of Participants; unit: Participants
Arm/Group | Personalized Therapy
Number analyzed (Participants) | 3
Participants | 0

ADVERSE EVENTS:
Time Frame: From the time the participant signs the informed consent until the study was stopped, an average of 16 months
Arm/Group | Personalized Therapy
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Personalized Therapy (N=3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anaphylaxis (Immune system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine increased (Investigations) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (3)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (3)
Fatigue (General disorders) | 2 (3)
Fever (General disorders) | 2 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized edema (General disorders) | 1 (1)
Gastrointestinal disorders-other, black stool (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Herpes simplex reactivation (Infections and infestations) | 1 (1)
Hotflashes (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Musculoskeletal and connective tissue disorders-other, body aches (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (6)
Non-cardiac chest pain (General disorders) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Papulopustular (Infections and infestations) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 2 (2)
Rash pustular (Infections and infestations) | 1 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-11): https://cdn.clinicaltrials.gov/large-docs/12/NCT02560012/Prot_SAP_000.pdf